CLINICAL TRIAL: NCT01276821
Title: Efficacy of Nebulised Hypertonic Saline (3%) Among Children With Mild to Moderately Severe Bronchiolitis - A Double Blind Randomized Controlled Trial.
Brief Title: Efficacy of Nebulised Hypertonic Saline (3%) Among Children With Bronchiolitis.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Aayush Khanal, MD (Other)
Responsible Party: Sponsor-Investigator, Dr. Aayush Khanal, MD, MD, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Organization: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEDSTUTHIOM
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Results first posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-04

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; L-Epinephrine; 3% Hypertonic Saline; Clinical Severity Score
MeSH Terms: conditions — Bronchiolitis | interventions — Saline Solution; Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Treatment (Placebo Comparator): L-Epinephrine and Normal Saline (0.9%)
  Interventions: Drug: L-Epinephrine and Normal Saline (0.9%)
- Study Treatment (Active Comparator): L-Epinephrine and Hypertonic Saline (3%)
  Interventions: Drug: L-Epinephrine and Hypertonic Saline (3%)

INTERVENTIONS:
Drug: L-Epinephrine and Normal Saline (0.9%) — 1.5ml of 1:1,000 L-Epinephrine and 4 ml of 0.9% Normal Saline
  Other Names: Nebulised Epinephrine in 0.9% Normal saline
  Arms: Standard Treatment
Drug: L-Epinephrine and Hypertonic Saline (3%) — 1.5ml of 1:1,000 L-Epinephrine and 4 ml of 3% Hypertonic Saline
  Other Names: Nebulised Epinephrine in 3% Hypertonic Saline
  Arms: Study Treatment

SUMMARY:
To assess the efficacy of nebulized 3% hypertonic saline in improving clinical severity scores among children aged 6 weeks to 24 months with bronchiolitis.

DETAILED DESCRIPTION:
Introduction and Rationale:

Bronchiolitis is a common problem with significant morbidity, and occasional mortality among young infants. Diagnostic testing, indications for hospitalization, eligibility criteria for discharge and therefore, the length of hospital stay for bronchiolitis vary globally, suggesting a lack of consensus and an opportunity to improve care for this common disorder. Likewise, despite the frequency of this condition there is no single, widely practiced, evidence-driven and universally accepted therapeutic guidelines other than supportive care. Recent studies have shown promising results regarding the role of nebulised 3% hypertonic saline in the treatment of bronchiolitis.

This therapy might obviate the need for hospital admission and reduce the length of hospital stay, if found effective. The implications of this would be that children return home early and parents return to work earlier, resulting in reduction of the morbidity and cost associated with the disease.

Trial Design This study was a prospective, interventional, parallel-assigned, double-blind, (subject,caregiver, investigator, outcome assessor) randomized controlled trial.

Ethical Clearance The study was approved by Institutional Review Board and Ethics Committee, Tribhuvan University Teaching Hospital, Institute of Medicine as well as The Institutional Review Board of Kanti Children's Hospital.

Study Participants Subjects were recruited from previously healthy children aged 6 weeks to 24 months visiting the Emergency Room and Out-Patient Department of Kanti Children Hospital with first episode of bronchiolitis.

Bronchiolitis was clinically defined as per the AAP consensus guidelines as the first episode of acute wheezing in children less than two years of age, starting as a viral upper respiratory infection (coryza, cough or fever).

Study setting The study was carried out in the Emergency Room, Observation and Out-Patient Department of Kanti Children Hospital, Kathmandu, Nepal. Recruitment occurred at the peak of bronchiolitis season in between January 15th to April 15th for duration of 4 months.

Interventions Patient enrollment occurred on weekdays (Sunday to Friday) between approximately 08.00 and 17.00 hr when, after the initial assessment, the attending pediatrician (non-study physician) called the investigator. The investigator assessed the children for eligibility, examined the children and assigned a clinical severity score described by Wang et al.

Children meeting inclusion criteria were invited to participate in the study and written informed consent was obtained from a parent or guardian.

General condition, weight, temperature, respiratory rate, heart rate, SpO2 and presence/absence of clinical dehydration were assessed in all patients and Clinical Severity score was calculated as described by Wang et al. Patients determined to be in life threatening condition were immediately managed for same and were not further considered for study.

Preparation of study drugs was done by a faculty appointed by the Department of Child Health and administration was done by an ER/OPD nurse or the investigator, and compliance with medication administration was assured by the investigator's direct observation of each nebulization.

All eligible patients were randomly assigned to one of the two groups:

1. Group 1 (n = 50) received inhalation of L-Epinephrine 1.5 mg, diluted to 4ml with 3% Hypertonic Saline (HS) solution;
2. Group 2 (n=50) received inhalation of L-Epinephrine, 1.5 mg, diluted to 4ml with 0.9% Normal Saline solution.

The study drug was administered at 0 and 30 min by jet nebulizers using a face mask. Prior to each drug administration and at 30, 60 and 120 min, the investigator assessed the children's general condition and recorded the CS score, SpO2 in room air, respiratory rate 60 and heart rate. All patients received the first dose of nebulization within 15- 30 minutes depending upon the time required for preparation and enrollment.

Adverse events were defined as heart rate >200, tremor, withdrawal from the study due to worsening clinical status, or discontinuation of any study medications due to side effects.

Patients were excluded from the study if the administration of the 2 courses of nebulisation was not delivered, the study drug was delayed by 10 min or more (protocol deviation) or if clinical deterioration mandated escalation of therapy and/or support.

At the end of the observation period, the attending pediatrician determined the need for hospital admission.

The parents of the patients enrolled in the study were asked to follow up after 24 hours in the OPD for repeat assessment. If the parents were not available for follow up, the investigator contacted the parents or guardians via telephone 24 hours after their ED/OPD discharge to determine the need for any unscheduled hospital visit within the next 24 hours of OPD/ ER visit: their readmission (relapse) rate.In addition, they were reassessed at the end of 1 week by telephone contact . A single investigator participated in the measurement of observations to minimize inter observer variability. All calls were made from the Hospital reception Office at appropriate times 10:00a.m. - 14:00p.m NST. Patient were labeled as Lost-to-Follow up if there was failure to communicate for 3 consecutive attempts for 2 consecutive days at their 7th and 8th day of initial presentation to the OPD/ER.

Sample Size Estimation:

Sample size was determined by the following formula :

* n = [(z1 +z2)² (Ó1² + Ó2²) ] / (û1 - û2)²
* Allowing a Type1 error of 5% (α :0.05), z1 score : 1.96.
* For a Power of 95%, z2=1.64.
* Standard deviation of the Clinical Severity Score : 1.3
* Mean Change in Clinical Severity Score between the two interventions to consider clinically significant : Change in Clinical Severity Score of 1
* The study proposed that a difference of 1 point in the Clinical Severity Score between the two intervention groups would be considered Clinically Significant.
* To detect this mean difference of 1 unit in the Clinical severity score, with a Power of 95%, a Sample size of 44 in each intervention group were required.This made a total of 88 patients to be enrolled in the study.Considering the drop out/ lost to follow up to be approximately 10%, 100 patients were enrolled, allowing 50 in each group.
* Standard deviation of the Change in clinical severity score was derived from previous studies and taken as 1.3 .

Randomization

1. Sequence Generation A Random Allocation Software generated by computer, identified patients by a triple digit mixed numeric code was used by the study coordinator to allocate patients to treatment groups, and the study coordinator was the only person with access to the randomization.
2. Type of Randomization Block Randomization method was used to stratify patients into blocks of 10 each, each comprising of 10 patients.

Allocation Concealment After preparation, the study solutions were labeled with the codes and wrapped in an envelope with the respective codes and attached with the proforma bearing the respective codes.Study solutions were identical in appearance and odor. The identity of the study solutions was blinded to all participants, care providers, and investigators and outcome assessor.

Implementation The randomization process was done by the study coordinator (not involved in the study) and he was the only person to have access to the codes.

The study solutions were stored in the non-freezer compartment of the refrigerator at a temperature of 2-8*C and were discarded if not used within 72 hours of preparation.

Blinding The study was a Double Blind Randomized Controlled Trial with the investigator, the participants, the nurses who delivered the drug, and the outcome assessor being blinded to the therapeutic option.

Statistical Methods The primary outcome was to detect the difference in mean change in Clinical Severity score between the two intervention groups. A power analysis revealed that, for detection of the difference of 1 unit in CS score between the 2 treatment groups, with α of 0.05 and power of 95%, we required 88 patients (44 per group).

A sample size of 100 patients was therefore chosen, with 50 patients in each group considering the possibility of loss to follow up.

Statistical analysis was performed using SPSS for Windows, Release 16.0 (SPSS Inc., Chicago, IL). Dichotomous events were analyzed by using the Chi-Square test.Dependent variables were compared by Student t-test. Statistical significance was defined as p-value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 weeks to 24 Months.
* First episode of wheezing
* Fever, cough and watery nasal discharge

Exclusion Criteria :

* Any underlying cardiovascular disease.
* Prior wheezing.
* Clinical Severity Score > 9.
* Atopic dermatitis, allergic rhinitis or asthma.
* Oxygen saturation (SpO2) <85% on room air.
* Obtunded consciousness.
* Previous treatment with bronchodilators within 4 hours.
* Any steroid therapy within 48 Hours.

Ages: 6 Weeks to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aayush Khanal, MD, Principal Investigator — Department of Child Health , Institute of Medicine , Tribhuvan University Teaching Hospital.; Arun Sharma, MD, Study Director — Department of Child Health , Tribhuvan University Teaching Hospital , Institute of Medicine, Maharajgunj, Kathmandu ,Nepal.; Srijana Basnet, MD, Study Director — Department of Child Health , Tribhuvan University Teaching Hospital , Institute of Medicine , Maharajgunj , Kathmandu , Nepal.; Pushpa R Sharma, DCH,FCPS, Study Chair — Head of the Department. Department of Child Health , Tribhuvan University Teaching Hospital , Institute of Medicine , Maharajgunj , Kathmandu , Nepal.; Fakir C Gami, MD, Study Chair — Department of Child Health, Tribhuvan University Teaching Hospital, Institute of Medicine.
Locations (1):
- Out Patient Department and Emergency Department, Kanti Children Hospital, Kathmandu, Bagmati Zone, Nepal

REFERENCES:
- [Derived] Khanal A, Sharma A, Basnet S, Sharma PR, Gami FC. Nebulised hypertonic saline (3%) among children with mild to moderately severe bronchiolitis--a double blind randomized controlled trial. BMC Pediatr. 2015 Sep 10;15:115. doi: 10.1186/s12887-015-0434-4. PMID 26357896

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from previously healthy children aged 6 weeks to 24 months with first episode of wheezing who visited the OPD and ER of Kanti Children Hospital and met the clinical definition of bronchiolitis.
  Recruitment occurred on weekdays from 8:00 to 17:00 Hours. Out of 754 screened children, 159 were first episode wheezers.
Groups:
- Standard: Nebulisation with 4ml of 0.9% Normal Saline and 1.5ml of L-Epinephrine
- Study: Nebulisation with 4ml of Hypertonic Saline (3%) and 1.5ml of L-Epinephrine
Period: Overall Study
Arm/Group | Standard | Study
Started | 50 | 50
Completed | 50 | 49
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard | Study | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 50 | 100
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: months] | 9.82 (5.06) | 9.51 (4.28) | 9.66 (4.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 23 | 52
  Male | 21 | 27 | 48
Region of Enrollment [Number; unit: participants]
  Nepal | 50 | 50 | 100
Duration of illness (days) [Mean (Standard Deviation); unit: Days] | 3.33 (0.96) | 3.43 (1.02) | 3.38 (0.99)
Clinical Severity Score Units [Mean (Standard Deviation); unit: Clinical Severity Score Units] — The Clinical Severity scoring system initially described by Wang, assesses respiratory rate, wheezing, retraction, and general condition,to assess the degree of respiratory distress in young children. It provides a score ranging from 0 to 12, with increased severity receiving a higher score.
  These scoring systems have previously been validated in a number of well designed randomized controlled trials (Anil 2010, Kuzik 2007, Sarrell 2002, and Mandelberg 2003). A 1 point improvement in the clinical severity score implies approximately 7% betterment of symptoms on the scale.
  Clinical Severity Score Units | 5.2 (1.1) | 5.3 (1.6) | 5.25 (1.35)
Respiratory Rate [Mean (Standard Deviation); unit: Breaths per minute] | 49 (2) | 49.1 (2.5) | 49.05 (2.25)
Spo2 (Oxygen Saturation) [Mean (Standard Deviation); unit: Percentage of Oxygen Saturation] | 93.5 (0.7) | 93.4 (0.8) | 93.45 (0.75)
Heart rate [Mean (Standard Deviation); unit: Beats per minute] | 149.7 (7.1) | 148.7 (7.5) | 149.2 (7.3)
Temperature [Mean (Standard Deviation); unit: Degrees Fahreinheit] | 99.2 (0.6) | 99.1 (0.6) | 99.15 (0.6)
Family History of Asthma, [Number; unit: participants]
  Positive | 5 | 4 | 9
  Negative | 45 | 46 | 91
Parental Smoking [Number; unit: participants] — History of parental Smoking (Secondhand passive smoke exposure status) of children
  participants
    Yes | 21 | 30 | 51
    No | 29 | 20 | 49
Enrollment from Emergency Department [Number; unit: participants]
  Enrollment from Emergency Room | 2 | 2 | 4
  Enrollment from Out-Patient Department | 48 | 48 | 96
Exposure to Biofuels [Number; unit: participants]
  Yes | 8 | 14 | 22
  No | 42 | 36 | 78
Breastfeeding Status [Number; unit: participants]
  Yes | 48 | 48 | 96
  No | 2 | 2 | 4
Prematurity [Number; unit: participants]
  Yes | 2 | 3 | 5
  No | 48 | 47 | 95
History suggestive of Atopy [Number; unit: participants]
  Yes | 3 | 7 | 10
  No | 47 | 43 | 90

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Clinical Severity Score
Description: Mean changes in the Clinical Severity Score after 2 sessions of nebulisation as compared to baseline.
  Clinical Severity Score devised by Wang et al, is an objective scoring system that measures the degree of respiratory distress in young children.
  The scoring system assesses respiratory rate, wheezing, retraction, and general condition,scores ranging from 0 to 3, with higher scores indicating severe illness and vice versa.
  The total scores range from 0 to 12, with increased severity receiving a higher score (Wang et al, 1992).
  This scoring systems have previously been validated in a number of well designed randomized controlled trials(Anil 2010, Kuzik 2007, Sarrell 2002, and Mandelberg 2003). A 1 point improvement in the clinical severity score implies approximately 7% betterment of symptoms on the scale.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard | Study
Number analyzed (Participants) | 50 | 50
units on a scale | 2.26 (1.15) | 3.57 (1.41)
Statistical Analysis 1: Comparison: Standard vs Study; Null Hypothesis Efficacy of nebulised hypertonic saline (3%) with L-Epinephrine is not higer than as compared to L-Epinephrine given with 0.9% normal saline in the management of children aged 6 weeks to 24 months with mild to moderately severe bronchiolitis. Alternate Hypothesis: Nebulised hypertonic saline (3%) with L-Epinephrine is superior to 0.9% Normal saline with L-Epinephrine in the management of children aged 6 weeks to 24 months with mild to moderately severe bronchiolitis; Test type: Non-Inferiority or Equivalence — Non - Inferiority Analysis; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 1.33, 95% CI 2-sided [0.78 to 1.82], Standard Deviation 1.30

2. Secondary Outcome: Patients Meeting Eligibility Criteria for ER/ OPD Discharge at the End of 2 Hours of Observation
Time Frame: At the end of 2 hours
Measure: Number; unit: participants
Arm/Group | Standard | Study
Number analyzed (Participants) | 50 | 50
participants
  Meets Criteria for ER/OPD discharge after 120 mins | 15 | 35
  Does not meet criteria for ER/OPD discharge | 35 | 15

3. Secondary Outcome: Relapse Rate
Description: To study the number of patients in either group who need another unscheduled medical visit within the initial 24 hours of ER/ OPD visit
Time Frame: 24 hours
Measure: Number; unit: Participants
Arm/Group | Standard | Study
Number analyzed (Participants) | 50 | 50
Participants
  Hospital Re-visit within 24 hours | 15 | 5
  No Hospital Re-visit within 24 hours | 35 | 45

4. Secondary Outcome: Need for Unscheduled Medical Visits, if Any, for Same Symptoms to Any Healthcare Facility Within 1 Week
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Standard | Study
Number analyzed (Participants) | 50 | 50
participants
  Unscheduled medical Visits in 1 week | 23 | 18
  No Unscheduled medical visits in 1 week | 27 | 32

5. Secondary Outcome: Missed Days of Work of Caregivers
Description: Number of patients in each intervention group whose parents reported at least 1 day of missed work due to the illness of child within the week following the initial hospital visit on 7 day follow-up call.
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Standard | Study
Number analyzed (Participants) | 50 | 50
participants | 10 | 3

6. Secondary Outcome: Persistence of Cough at the End of 1 Week
Description: Number of patients in each intervention group whose parents reported the persistence of initial cough at the end of 1 week in their children.
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Standard | Study
Number analyzed (Participants) | 50 | 50
participants
  Persistence of cough at the end of 1 week | 37 | 31
  Absence of cough at the end of 1 week | 13 | 19

7. Other Pre Specified Outcome: Average Duration of Crying (in Minutes) Among Babies Receiving Nebulisation Therapy.
Description: The outcomes tries to compare the influence of duration of crying among babies receiving nebulization which interferes with drug delivery and henceforth might create a confounding bias while interpreting results.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Standard | Study
Number analyzed (Participants) | 50 | 50
Minutes | 2.16 (0.79) | 2.03 (0.90)

ADVERSE EVENTS:
Arm/Group | Standard | Study
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes